CLINICAL TRIAL: NCT00257465
Title: M-Vax: A Feasibility and Bio-Equivalence Study Using a DNP-Modified Autologous Melanoma Tumor Cell Vaccine as Therapy in Patients With Stage III or IV Melanoma
Brief Title: Trial of Autologous, Hapten-Modified Vaccine in Patients With Stage III or IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AVAX Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A/100/0401
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma
Keywords: melanoma; metastatic; vaccine; immunotherapy; autologous
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): 'Autologous, DNP-modified vaccine (M-Vax)'
  Interventions: Biological: Autologous, DNP-modified vaccine (M-Vax); Biological: Autologous, DNP-Modified Melanoma Vaccine
- B (Experimental): Autologous, DNP-Modified Vaccine (MVax)
  Interventions: Biological: Autologous, DNP-modified vaccine (M-Vax); Biological: Autologous, DNP-Modified Vaccine
- C (Experimental): Autologous, DNP-Modified Vaccine (MVax)
  Interventions: Biological: Autologous, DNP-modified vaccine (M-Vax); Biological: Autologous, DNP-Modified Vaccine
- D (Placebo Comparator): 0 cells
  Interventions: Biological: Autologous, DNP-Modified Vaccine

INTERVENTIONS:
Biological: Autologous, DNP-modified vaccine (M-Vax) — 5.0, 2.5, 0.5, or 0 cells
  Arms: A; B; C
Biological: Autologous, DNP-Modified Melanoma Vaccine — 5 million cells
  Other Names: MVax
  Arms: A
Biological: Autologous, DNP-Modified Vaccine — 2.5 million cells
  Other Names: MVax
  Arms: B
Biological: Autologous, DNP-Modified Vaccine — 0.5 million cells
  Other Names: MVax
  Arms: C
Biological: Autologous, DNP-Modified Vaccine — 0 cells
  Other Names: MVax
  Arms: D

SUMMARY:
The purpose of this study is to determine whether a vaccine composed of patients' own melanoma cells treated with the chemical, dinitrophenyl (DNP)(called a hapten), is safe and stimulates an immune response to patients' own cancer cells.

DETAILED DESCRIPTION:
Patients with stage III or IV melanoma need to have at least one tumor mass of at least 2.5 cm (about 1 inch) diameter than can be removed for vaccine production. If the vaccine is successfully made and if the patient is eligible, the patient will be assigned to receive one of 4 doses of the vaccine, include one group that will receive a zero dose. All patients will receive injections of their vaccine as part of immune system testing and will receive low dose cyclophosphamide and BCG. Eight injections of the vaccine will be administered as an injection into the skin of the arm over a 6 month period. Before and after vaccine administration, patients will be tested for immunity to their own melanoma cells by DTH testing, which is similar to a tuberculosis test. All side effects caused by the vaccine will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* stage III or IV melanoma at least one tumor mass of at least 2.5 cm diameter that can be excised to make vaccine good performance status

Exclusion Criteria:

* brain metastases need for steroids or other immunosuppressive drugs positive PPD tests positive test for HIV, hepatitis B (antigen), or hepatitis C other serious medical illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Immune response to patients' own melanoma cells | 2 months

SECONDARY OUTCOMES:
Safety | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: David Berd, MD, Principal Investigator — AVAX Technologies
Locations (7):
- United States (7):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Pacific Oncology and Hematology Associates, San Diego, California
  - University of Illinois School of Medicine, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Berd D, Sato T, Maguire HC Jr, Kairys J, Mastrangelo MJ. Immunopharmacologic analysis of an autologous, hapten-modified human melanoma vaccine. J Clin Oncol. 2004 Feb 1;22(3):403-15. doi: 10.1200/JCO.2004.06.043. Epub 2003 Dec 22. PMID 14691123